CLINICAL TRIAL: NCT06272240
Title: Study of the Role of the Tumor Microenvironment in Ovarian Cancer
Brief Title: Tumor Microenvironment in Ovarian Cancer
Acronym: MICO
Status: Recruiting | Type: Observational
Sponsor: University of Udine (Other)
Responsible Party: Sponsor
Other Study IDs: 17380
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer Stage III; Ovarian Cancer Stage IV
Keywords: organoids,tumor microenviroment,ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Patients with primary diagnosis (t=0) of epithelial ovarian cancer (stage III and IV according to FIGO) cadidate for surgical removal will be selected. The removed tissue will be sent to the Pathology Department, where it will be selected by the pathologist, who will collect a fragment of tumor tissue and one from adjacent normal tissue (as a healthy control) and will divide them into three parts: one for the identification of cells composing the Tumor Microenvironment (TME) (through single-cell analysis), one for microbiome analysis, and one for organoid generation to be conducted at the laboratories of the Department of Medical Area.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ovarian Cancer Organoids — To characterize in vitro interactions and molecular pathway among tumor cells, immune cells, and resident microbiota (intratumoral bacteria and/or microbial-derived molecules)

SUMMARY:
A detailed understanding of molecular mechanism of cancer genesis is fundamental to develop innovative and personalized therapies. The new frontier in biomedical research is represented by organoids, a three-dimensional cell culture system obtained from a tissue fragment that accurately reproduces the essential properties of the original tissue in vitro, which could provide a valuable model for explanation of ovarian cancers pathogenesis and will allow to predict the response to a specific therapy. With this research project, we expect to generate ovarian cancer organoids to characterize in vitro interactions and molecular pathway among tumor cells, immune cells, and resident microbiota (intratumoral bacteria and/or microbial-derived molecules).

DETAILED DESCRIPTION:
Background Proved the importance of microenviroment in the onset and progression of ovarian cancer, a detailed understanding of molecular mechanism of cancer genesis is fundamental to develop innovative and personalized therapies.

Primary Objective The new frontier in biomedical research is represented by organoids, a three-dimensional cell culture system obtained from a tissue fragment that accurately reproduces the essential properties of the original tissue in vitro, which could provide a valuable model for explanation of ovarian cancers pathogenesis and will allow to predict the response to a specific therapy.

Study Hypothesis To generate of ovarian cancer organoids to characterize in vitro interactions and molecular pathway among tumor cells, immune cells, and resident microbiota (intratumoral bacteria and/or microbial-derived molecules).

Trial Design Patients with primary diagnosis of epithelial ovarian cancer (EOC) (stage III and IV according to FIGO) referred to the Obstetrics-Gynecology Department of ASUFC for surgical removal will be selected. It is expected that organoids will be cultured from 50 patients over the course of 3 years, obtained by removed tissue from which pathologist will collect a fragment of tumor tissue and one from adjacent normal tissue (as a healthy control). From tumor tissue they will extract three different fragments: one for the identification of cells composing the Tumor Microenvironment (TME) (through single-cell analysis), one for microbiome analysis, and one for organoid generation to be conducted at the laboratories of the Department of Medical Area.

Inclusion/Exclusion Criteria Patients with a diagnosis of EOC will be considered eligible if they meet these criteria: Age: 18 years - 80 years, serous ovarian carcinoma and FIGO Stage III/IV EOC. They will be excluded in case of ongoing or suspended immunosuppressive therapy within the last 6 months, congenital or acquired immunodeficiency, immunosuppressive state, administration of chemotherapy for another neoplasm in the past 12 months, non-epithelial ovarian tumors, patients not undergoing surgical intervention, BMI higher than 30, absence of Informed Consent.

Primary Endpoint With this research project, we expect to understand if it is also possible to stratify ovarian cancer patients based on the activation of AhR in cells of the Tumor Microenvironment (TME), including tumor cells and immune cells.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Age < 80 years
* Serous ovarian carcinoma
* FIGO Stage III-IV

Exclusion Criteria:

* Ongoing or suspended immunosuppressive therapy within the last 6 months
* Congenital or acquired immunodeficiency
* Immunosuppressive state
* Administration of chemotherapy for another neoplasm in the past 12 months
* Non-epithelial ovarian tumors
* Patients not undergoing surgical intervention
* BMI > 30
* Absence of Informed Consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with primary diagnosis (t=0) of epithelial ovarian cancer (stage III and IV according to FIGO)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
• Composition of the tumor microenvironment (including the immune system and intratumoral microbiota). • Generate organoids | from enrollment to the end of follow up at 36 months
  Characterize the composition of the tumor microenvironment (including the immune system and intratumoral microbiota). Generate organoids from cells derived from ovarian tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Udine, Udine, UD, Italy

REFERENCES:
- [Background] Nejman D, Livyatan I, Fuks G, Gavert N, Zwang Y, Geller LT, Rotter-Maskowitz A, Weiser R, Mallel G, Gigi E, Meltser A, Douglas GM, Kamer I, Gopalakrishnan V, Dadosh T, Levin-Zaidman S, Avnet S, Atlan T, Cooper ZA, Arora R, Cogdill AP, Khan MAW, Ologun G, Bussi Y, Weinberger A, Lotan-Pompan M, Golani O, Perry G, Rokah M, Bahar-Shany K, Rozeman EA, Blank CU, Ronai A, Shaoul R, Amit A, Dorfman T, Kremer R, Cohen ZR, Harnof S, Siegal T, Yehuda-Shnaidman E, Gal-Yam EN, Shapira H, Baldini N, Langille MGI, Ben-Nun A, Kaufman B, Nissan A, Golan T, Dadiani M, Levanon K, Bar J, Yust-Katz S, Barshack I, Peeper DS, Raz DJ, Segal E, Wargo JA, Sandbank J, Shental N, Straussman R. The human tumor microbiome is composed of tumor type-specific intracellular bacteria. Science. 2020 May 29;368(6494):973-980. doi: 10.1126/science.aay9189. PMID 32467386
- [Background] Banerjee S, Tian T, Wei Z, Shih N, Feldman MD, Alwine JC, Coukos G, Robertson ES. The ovarian cancer oncobiome. Oncotarget. 2017 May 30;8(22):36225-36245. doi: 10.18632/oncotarget.16717. PMID 28410234
- [Background] Yang J, Huang S, Cheng S, Jin Y, Zhang N, Wang Y. Application of Ovarian Cancer Organoids in Precision Medicine: Key Challenges and Current Opportunities. Front Cell Dev Biol. 2021 Aug 2;9:701429. doi: 10.3389/fcell.2021.701429. eCollection 2021. PMID 34409036
- [Background] Ranhotra HS, Flannigan KL, Brave M, Mukherjee S, Lukin DJ, Hirota SA, Mani S. Xenobiotic Receptor-Mediated Regulation of Intestinal Barrier Function and Innate Immunity. Nucl Receptor Res. 2016;3:101199. doi: 10.11131/2016/101199. PMID 27942535
- [Background] Hezaveh K, Shinde RS, Klotgen A, Halaby MJ, Lamorte S, Ciudad MT, Quevedo R, Neufeld L, Liu ZQ, Jin R, Grunwald BT, Foerster EG, Chaharlangi D, Guo M, Makhijani P, Zhang X, Pugh TJ, Pinto DM, Co IL, McGuigan AP, Jang GH, Khokha R, Ohashi PS, O'Kane GM, Gallinger S, Navarre WW, Maughan H, Philpott DJ, Brooks DG, McGaha TL. Tryptophan-derived microbial metabolites activate the aryl hydrocarbon receptor in tumor-associated macrophages to suppress anti-tumor immunity. Immunity. 2022 Feb 8;55(2):324-340.e8. doi: 10.1016/j.immuni.2022.01.006. PMID 35139353
- [Background] Tuveson D, Clevers H. Cancer modeling meets human organoid technology. Science. 2019 Jun 7;364(6444):952-955. doi: 10.1126/science.aaw6985. PMID 31171691
- [Background] Ricci F, Bizzaro F, Cesca M, Guffanti F, Ganzinelli M, Decio A, Ghilardi C, Perego P, Fruscio R, Buda A, Milani R, Ostano P, Chiorino G, Bani MR, Damia G, Giavazzi R. Patient-derived ovarian tumor xenografts recapitulate human clinicopathology and genetic alterations. Cancer Res. 2014 Dec 1;74(23):6980-90. doi: 10.1158/0008-5472.CAN-14-0274. Epub 2014 Oct 10. PMID 25304260
- [Derived] Arcieri M, Capezzali E, Restaino S, Pregnolato S, Mariuzzi L, Mangogna A, Orsaria M, Tulisso A, Tonon S, De Martino M, Isola M, Driul L, Pucillo C, Scambia G, Frossi B, Vizzielli G. Study of the Role of the Tumor Microenvironment in Ovarian Cancer (MICO): A Prospective Monocentric Trial. Cancer Rep (Hoboken). 2025 Jun;8(6):e70242. doi: 10.1002/cnr2.70242. PMID 40464605